CLINICAL TRIAL: NCT05050097
Title: A Multi-arm Phase 1b Study of Talquetamab With Other Anticancer Therapies in Participants With Multiple Myeloma
Brief Title: A Study of Talquetamab With Other Anticancer Therapies in Participants With Multiple Myeloma
Acronym: MonumenTAL-2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108946; 64407564MMY1004 (Other: Janssen Research & Development, LLC); 2020-004502-55 (EudraCT Number); 2023-503620-60-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab; carfilzomib; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Regimen A: Talquetamab + Carfilzomib (Experimental): Participants assigned to Treatment regimen A will receive talquetamab subcutaneously (SC) in combination with carfilzomib as an intravenous (IV) infusion.
  Interventions: Drug: Talquetamab; Drug: Carfilzomib
- Treatment Regimen B: Talquetamab + Daratumumab + Carfilzomib (Experimental): Participants assigned to Treatment regimen B will receive talquetamab SC in combination with daratumumab SC and carfilzomib as an IV infusion.
  Interventions: Drug: Talquetamab; Drug: Carfilzomib; Drug: Daratumumab SC
- Treatment Regimen C: Talquetamab + Lenalidomide (Experimental): Participants assigned to Treatment regimen C will receive talquetamab SC in combination with lenalidomide orally.
  Interventions: Drug: Talquetamab; Drug: Lenalidomide
- Treatment Regimen D: Talquetamab + Daratumumab + Lenalidomide (Experimental): Participants assigned to Treatment regimen D will receive talquetamab SC in combination with daratumumab SC and lenalidomide orally.
  Interventions: Drug: Talquetamab; Drug: Daratumumab SC; Drug: Lenalidomide
- Treatment Regimen E: Talquetamab + Pomalidomide (Experimental): Participants assigned to Treatment regimen E will receive talquetamab SC in combination with pomalidomide orally.
  Interventions: Drug: Talquetamab; Drug: Pomalidomide

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564
Drug: Carfilzomib — Carfilzomib will be administered as an IV infusion.
  Arms: Treatment Regimen A: Talquetamab + Carfilzomib; Treatment Regimen B: Talquetamab + Daratumumab + Carfilzomib
Drug: Daratumumab SC — Daratumumab will be administered subcutaneously.
  Arms: Treatment Regimen B: Talquetamab + Daratumumab + Carfilzomib; Treatment Regimen D: Talquetamab + Daratumumab + Lenalidomide
Drug: Lenalidomide — Lenalidomide will be self-administered orally.
  Arms: Treatment Regimen C: Talquetamab + Lenalidomide; Treatment Regimen D: Talquetamab + Daratumumab + Lenalidomide
Drug: Pomalidomide — Pomalidomide will be self-administered orally.
  Arms: Treatment Regimen E: Talquetamab + Pomalidomide

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of talquetamab when administered in different combination regimens and to identify the safe dose(s) of talquetamab combination regimens.

ELIGIBILITY:
Inclusion Criteria:

* Have documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Have measurable disease at screening as defined by at least 1 of the following: a. Serum monoclonal protein (M-protein) level greater than or equal to (>=) 1.0 gram per deciliter (g/dL); or b. Urine M-protein level >= 200 milligrams (mg)/24 hours; or c. Light chain multiple myeloma: Serum immunoglobulin (Ig) free light chain (FLC) >=10 milligrams per deciliter (mg/dL) and abnormal serum Ig kappa lambda FLC ratio
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 at screening and immediately before the start of study treatment administration
* A woman of childbearing potential must have a negative highly sensitive serum beta human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine or serum pregnancy test within 24 hours before the start of study treatment administration
* Be willing and able to adhere to the lifestyle restrictions specified in the protocol, including adherence to the applicable immunomodulatory drug (IMiD) global Pregnancy Prevention Plan (PPP) or local PPP/Risk Evaluation and Mitigation Strategy (REMS) program

Exclusion Criteria:

* Live, attenuated vaccine within 4 weeks before the first dose of study treatment
* Received a cumulative dose of corticosteroids equivalent to >=140 mg of prednisone within the 14-day period before the start of study treatment administration
* Active central nervous system (CNS) involvement or exhibition of clinical signs of meningeal involvement of multiple myeloma. If either is suspected, brain magnetic resonance imaging (MRI) and lumbar cytology are required
* Known to be seropositive for human immunodeficiency virus
* History of stroke or seizure within 6 months prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 1 year and 10 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 1 year and 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to AE.
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Up to 1 year and 6 months
  Number of participants with clinically significant abnormalities in laboratory parameters such as hematology and serum chemistry will be reported.
Number of Participants with Dose Limiting Toxicity (DLT) | Up to 49 days
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity of grade 3 or higher, clinical laboratory abnormalities, or hematologic toxicity.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 1 year and 10 months
  ORR is defined as the percentage of participants who achieve partial response (PR) or better according to the International Myeloma Working Group (IMWG) 2016 criteria. Response to treatment will be evaluated by the investigator based on IMWG criteria.
Very Good Partial Response (VGPR) or Better Response Rate | Up to 1 year and 10 months
  VGPR or better response rate is defined as the percentage of participants who achieve a VGPR or better response (stringent complete response [sCR] + complete response [CR] +VGPR) according to the IMWG 2016 criteria.
Complete Response (CR) or Better Response Rate | Up to 1 year and 10 months
  CR or better response rate is defined as the percentage of participants who achieve a CR or better response (sCR+CR) according to the IMWG 2016 criteria.
Stringent Complete Response (sCR) | Up to 1 year and 10 months
  sCR rate is defined as the percentage of participants who achieve an sCR according to the IMWG 2016 criteria.
Duration of Response | Up to 1 year and 10 months
  Duration of response is defined as time from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG 2016 criteria, or death due to disease progression, whichever occurs first.
Time to Response | Up to 1 year and 10 months
  Time to response is defined as the time between date of first dose of study treatment and the first efficacy evaluation at which the participant has met all criteria for PR or better.
Serum Concentration of Talquetamab | Up to 1 year and 10 months
  Serum samples will be analyzed to determine concentrations of talquetamab.
Serum Concentration of Daratumumab | Up to 1 year and 10 months
  Serum samples will be analyzed to determine concentrations of daratumumab for treatment regimens B and D.
Number of Participants with Anti-Drug Antibodies to Talquetamab | Up to 1 year and 10 months
  Number of participants with anti-drug antibodies to talquetamab will be reported.
Number of Participants with Anti-Drug Antibodies to Daratumumab | Up to 1 year and 10 months
  Number of participants with anti-drug antibodies to daratumumab will be reported for treatment regimens B and D.
Number of Participants with Anti-Drug Antibodies to Recombinant Human Hyaluronidase PH20 Enzyme (rHuPH20) | Up to 1 year and 10 months
  Number of participants with anti-drug antibodies to rHuPH20 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (31):
- United States (12):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - St Vincents Hospital Melbourne, Fitzroy
  - Alfred Health, Melbourne
  - Gold Coast University Hospital, Southport
  - Wollongong Hospital, Wollongong
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - UZA, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- France (4):
  - CHU Nantes, Nantes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- Netherlands (3):
  - UMCG, Groningen
  - Maastricht University Medical Centre, Maastricht
  - UMCU, Utrecht
- United Kingdom (4):
  - University College Hospital London, London
  - The Christie Nhs Foundation Trust, Manchester
  - Churchill Hospital, Oxford
  - The Royal Marsden NHS Trust Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency